CLINICAL TRIAL: NCT00128037
Title: A Phase II Trial of Pre-operative Chemoradiotherapy Followed by Surgical Resection in Pancoast Tumors: Initial Report of Japan Clinical Oncology Group Trial (JCOG 9806)
Brief Title: Trial of Pre-operative Chemoradiotherapy Followed by Surgical Resection in Pancoast Tumors (JCOG 9806)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCOG 9806; C000000031
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Neoplasm
Keywords: pulmonary neoplasm; preoperative chemoradiotherapy; surgical resection; superior sulcus tumor; chest wall invasion; mytomicin C; vindesine; cisplatin
MeSH Terms: conditions — Lung Neoplasms; Pancoast Syndrome | interventions — Mitomycin; Vindesine; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: mitomycin C, vindesine, cisplatin and radiotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the trimodality (concurrent chemoradiotherapy followed by surgical resection) approach in superior sulcus tumors.

DETAILED DESCRIPTION:
Pre-operative radiotherapy has long been the community standard in Pancoast, or superior sulcus tumor. However, both complete resection rate (-50%) and long-term survival (-30%) are poor and unchanged for 40 years. Concurrent chemoradiotherapy has been shown to be beneficial in unresectable stage III non-small cell cancer. Surgery after induction chemoradiotherapy thus is a promising treatment strategy, and in fact, SWOG reported favorable results of this trimodality approach in superior sulcus tumor. The current trial is a Japanese, cooperative, multi-center, prospective one to evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, pathologically documented non-small cell lung cancer (NSCLC)
* Invasion to the first rib or more superior chest wall
* Age: 15-74 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Ample organ function
* No prior chemo- or radiotherapy
* Signed informed consent

Exclusion Criteria:

* Metastasis to, or involvement of, mediastinal node (N2)
* Distant metastasis or dissemination to pleura/pericardium
* Active concomitant malignancy
* Unstable angina, recent myocardial infarction, heart failure
* Uncontrolled diabetes or hypertension
* Pregnant or lactating women
* Other severe complications

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1999-05; Study Completion 2006-02

PRIMARY OUTCOMES:
3-year survival rate

SECONDARY OUTCOMES:
complete resection rate
post-surgical morbidity/mortality
local control rate

CONTACTS AND LOCATIONS:
Overall Officials: Harubumi Kato, M.D., Ph.D., Study Chair — Tokyo Medical University
Locations (1):
- National Cancer Center, Chuo-ku, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.jcog.jp/